CLINICAL TRIAL: NCT00898794
Title: Influence of Bevacizumab and VEGF on Platelet Aggregation
Brief Title: Effect of Bevacizumab and VEGF on Platelet Clustering in Patients Who Are Receiving Bevacizumab for Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kantonsspital Graubuenden (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: KSGR-GR-01-07; CDR0000631252 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2011-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — Bevacizumab; Bleeding Time; Platelet Aggregation

INTERVENTIONS:
Biological: bevacizumab
Other: coagulation study
Other: laboratory biomarker analysis
Other: platelet aggregation test

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about the effect of bevacizumab and VEGF on platelet clustering.

PURPOSE: This research study is looking at the effect of bevacizumab and VEGF on platelet clustering in patients with cancer who are receiving bevacizumab.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the influence of bevacizumab on platelet aggregation in patients receiving bevacizumab for cancer.
* To determine the influence of VEGF on platelet aggregation.
* To determine the influence of VEGF or bevacizumab on cyclooxygenesis.
* To determine if the sequence of medication plays a role in platelet aggregation.

OUTLINE: Blood samples are collected before and after bevacizumab infusion. Samples are analyzed for measurements of platelet aggregation, coagulation parameters, and endothelial activation (e.g., fibrin fragment F1 and 2, thrombin and antithrombin complex, soluble P-selectin, Von Willebrand factor and factor VIII, tissue factor, and endothelin 1).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Receiving bevacizumab for cancer

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Influence of bevacizumab on platelet aggregation
Influence of VEGF on platelet aggregation
Influence of VEGF or bevacizumab on cyclooxygenesis
Correlation between medication sequence and platelet aggregation

CONTACTS AND LOCATIONS:
Overall Officials: Roger von Moos, MD, Principal Investigator — Kantonsspital Graubuenden
Locations (1):
- Kantonsspital Graubuenden, Chur, Switzerland